CLINICAL TRIAL: NCT01980225
Title: Randomized Controlled Trial Comparing the Implantation Rate of Vitrified-warmed Blastocysts With and Without Artificial Shrinkage Before Vitrification
Brief Title: Implantation Rate of Vitrified-warmed Collapsed Blastocysts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Reproductive Medicine, Belgium (Other)
Responsible Party: Principal Investigator, Lisbet Van Landuyt, klinisch embryoloog, Centre for Reproductive Medicine, Belgium
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VanLanduyt2013
Record Dates: First submitted 2013-10-28; First posted 2013-11-08 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Implantation Rate of Vitrified Blastocysts
Keywords: vitrification, blastocyst, artificial shrinkage, collapse
MeSH Terms: conditions — Unconsciousness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Collapse (Experimental): This arm includes the patients where laser-induced collapse (=artificial shrinkage) of all blastocysts is performed before vitrification
  Interventions: Procedure: Collapse
- control (No Intervention): This control arm includes the patients of which the blastocysts are vitrified without performing collapse

INTERVENTIONS:
Procedure: Collapse — inducing collapse (= artificial shrinkage) by applying 1 or 2 laser pulses between trophectoderm cells of the blastocyst to be vitrified
  Other Names: artificial shrinkage
  Arms: Collapse

SUMMARY:
In our centre, the implantation rate of frozen blastocysts (cryopreserved using vitrification)was 20,3% (Van Landuyt et al. 2011). This implantation rate is lower when compared to data from other observational studies. Retrospective studies have shown that artificial shrinkage of the blastocoelic cavity (also called collapse) and dehydration of the blastocyst just before vitrification can have a positive effect on the survival after warming. This collapse can be induced by using a laser. The study of Iwayama et al. 2010 has shown a similar survival rate but an increase in the implantation rate of collapsed blastocysts compared to non-collapsed blastocysts.

The aim of the study is to investigate the effect of artificial shrinkage by laser-induced collapse on the implantation potential of vitrified-warmed day 5 or day 6 blastocyst stage embryos in a prospective randomised controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* female age <39 years
* at least 1 blastocyst available for cryopreservation

Exclusion Criteria:

* sperm origin: testicular or epididymal sperm extraction
* IVM (in-vitro maturation) cycles
* PGD cycles (preimplantation genetic diagnosis)

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 270 (Actual)
Dates: Start 2011-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
implantation rate of the embryo in the first frozen transfer cycle | approximately 10 weeks after the first frozen embryo transfer
  patients are enrolled in the study at oocyte retrieval. When patient is not pregnant after fresh embryo transfer, she comes back to use the frozen embryos at least one month after the initial inclusion. After the frozen embryo transfer, poshCG is measured 14 days after transfer. Approximately 10 weeks after transfer, implantation rate of the frozen embryos is assessed. This is the number of intra-uterine gestational sacs seen on ultrasound on the number of embryos transferred

SECONDARY OUTCOMES:
survival rate of warmed blastocysts | 0-30 minutes
  this is the morphological assessment of survival of the blastocyst after warming
implantation rate per warmed blastocyst | approximately 10 weeks after first frozen transfer
  implantation rate of the transferred embryo per embryo initially warmed in that frozen transfer cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Lisbet Van Landuyt, MSc, Principal Investigator — Centre for Reproductive Medicine
Locations (1):
- Centre for Reproductive Medicine, Brussels, Belgium

REFERENCES:
- [Derived] Van Landuyt L, Polyzos NP, De Munck N, Blockeel C, Van de Velde H, Verheyen G. A prospective randomized controlled trial investigating the effect of artificial shrinkage (collapse) on the implantation potential of vitrified blastocysts. Hum Reprod. 2015 Nov;30(11):2509-18. doi: 10.1093/humrep/dev218. Epub 2015 Sep 12. PMID 26364080